CLINICAL TRIAL: NCT04163991
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Mechanistic Insight and Dosage Optimization Study of the Efficacy and Safety of VIB4920 in Patients With Rheumatoid Arthritis (RA)
Brief Title: A Study to Evaluate the Safety and Efficacy of VIB4920 in Participants With Rheumatoid Arthritis
Acronym: MIDORA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIB4920.P2.S3; 2019-003697-70 (EudraCT Number)
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; VIB4920; MEDI4920
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- VIB4920 1500 mg 4 Times (Experimental): Participants receive intravenous (IV) infusion of VIB4920 1500 mg on Days 1, 15, 29, and 57
  Interventions: Drug: VIB4920
- VIB4920 1500 mg Twice (Experimental): Participants receive IV infusion of VIB4920 1500 mg on Days 1 and 57, placebo on Days 15 and 29.
  Interventions: Drug: VIB4920; Drug: Placebo
- VIB4920 3000 mg Twice (Experimental): Participants receive IV infusion of VIB4920 3000 mg on Days 1 and 57, placebo on Days 15 and 29.
  Interventions: Drug: VIB4920; Drug: Placebo
- VIB4920 3000 mg Once (Experimental): Participants receive IV infusion of VIB4920 3000 mg on Day 1 and placebo on Days 15, 29, and 57.
  Interventions: Drug: VIB4920; Drug: Placebo
- Placebo (Placebo Comparator): Participants receive IV infusion of placebo matched to VIB4920 on Days 1, 15, 29, and 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIB4920 — liquid for IV infusion following dilution in normal saline
  Other Names: MEDI4920; dazodalibep
  Arms: VIB4920 1500 mg 4 Times; VIB4920 1500 mg Twice; VIB4920 3000 mg Once; VIB4920 3000 mg Twice
Drug: Placebo — 0.9% saline for IV infusion
  Arms: Placebo; VIB4920 1500 mg Twice; VIB4920 3000 mg Once; VIB4920 3000 mg Twice

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, and pharmacokinetics (PK) of VIB4920 (formerly MEDI4920) in adult participants with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The overall study period will be approximately 337 days. After a screening period of up to 28 days, the participants will be randomized in a 1:1:1:1:1 ratio to receive intravenous dose of VIB4920 and/or placebo in 5 cohorts. Participants are to be followed on their stable background anti-RA therapy at least through 12 weeks (Day 85), at which time rescue therapy may be instituted. All participants will be followed at least through the primary (interim) analysis (Day 113), and those who have not instituted rescue therapy will be followed through Day 309 to determine the duration of clinical response. The primary analysis will be after all participants have completed Day 113, and the final analysis will be after all participants have completed follow-up.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Principal Inclusion Criteria:

1. Male or female adults, >= 18 years of age at time of informed consent.
2. Diagnosed with RA according to the European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) 2010 criteria >= 6 months prior to screening.
3. Disease Activity Score in 28 Joints (DAS 28) using C-reactive Protein (DAS28-CRP) > 3.2 at screening with >= 4 tender joint count (TJC) and >= 4 swollen joint count (SJC) out of the 28 joints assessed for DAS28 present at screening and confirmed present at visit 2 prior to randomization.
4. Positive for rheumatoid factor (RF) and/or anti-citrullinated protein antibodies (ACPA) at screening, in accordance with criteria at the central laboratory.
5. Treated with methotrexate (MTX), with or without a concomitant conventional disease-modifying anti-rheumatic drug (cDMARD).
6. Agreeing to use of protocol defined contraception methods.

Principal Exclusion Criteria:

1. Prior or current inflammatory joint disease other than RA.
2. Severe interstitial lung disease.
3. Prior receipt of any biologic B-cell-depleting therapy.
4. Receipt of any anti - tumor necrosis factor alpha (TNF-α) biologic agent < 8 weeks prior to screening.
5. Receipt of any biologic disease-modifying anti-rheumatic drug (bDMARD) with a mechanism of action other than direct TNF-α blockade, < 12 weeks or < 5 half-lives of the drug prior to screening.
6. Injectable corticosteroids or treatment with > 10 mg/day dose of oral prednisolone or equivalent within 4 weeks prior to screening.
7. Previous treatment with anti-cluster of differentiation 40 ligand (CD40L) compounds at any time before randomization.
8. Hepatitis B, hepatitis C, or human immunodeficiency virus infection.
9. Pregnant or lactating or planning to get pregnant during the duration of the study.
10. Evidence of active tuberculosis (TB) or being at high risk for TB.
11. History of more than one episode of herpes zoster in the 12 months prior to screening or any opportunistic infection in the 12 months prior to screening, excluding localized mucocutaneous candidiasis.
12. Receipt of live vaccine or live therapeutic infectious agent within the 4 weeks prior to screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (25):
- United States (18):
  - Research Site, Anniston, Alabama
  - Research Site, Sun City, Arizona
  - Research Site, Upland, California
  - Research Site, Clearwater, Florida
  - Research Site, Margate, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Lexington, Kentucky
  - Research Site, Wheaton, Maryland
  - Research Site, Charlotte, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Vandalia, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Baytown, Texas
  - Research Site, Dallas, Texas
- Poland (7):
  - Research Site, Poznan, Greater Poland Voivodeship
  - Research Site, Krakow, Lesser Poland Voivodeship
  - Research Site, Nadarzyn, Masovian Voivodeship
  - Research Site, Siedlce, Masovian Voivodeship
  - Research Site, Bialystok, Podlaskie Voivodeship
  - Research Site, Elblag, Warmian-Masurian Voivodeship
  - Research Site, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kivitz A, Wang L, Alevizos I, Gunsior M, Falloon J, Illei G, St Clair EW. The MIDORA trial: a phase II, randomised, double-blind, placebo-controlled, mechanistic insight and dosage optimisation study of the efficacy and safety of dazodalibep in patients with rheumatoid arthritis. RMD Open. 2023 Aug;9(3):e003317. doi: 10.1136/rmdopen-2023-003317. PMID 37541743

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a screening period of up to 28 days, eligible participants were randomized in a 1:1:1:1:1 ratio into 5 cohorts.
Groups:
- Placebo: Participants received intravenous (IV) infusion of placebo matched to VIB4920 on Days 1, 15, 29, and 57.
- VIB4920 3000 mg Once: Participants received IV infusion of VIB4920 3000 mg on Day 1 and placebo on Days 15, 29, and 57.
- VIB4920 1500 mg Twice: Participants received IV infusion of VIB4920 1500 mg on Days 1 and 57, placebo on Days 15 and 29.
- VIB4920 3000 mg Twice: Participants received IV infusion of VIB4920 3000 mg on Days 1 and 57, placebo on Days 15 and 29.
- VIB4920 1500 mg 4 Times: Participants received IV infusion of VIB4920 1500 mg on Days 1, 15, 29, and 57.
Period: Overall Study
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Started | 16 | 16 | 16 | 15 | 15
Completed | 15 | 13 | 11 | 12 | 14
Not Completed | 1 | 3 | 5 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 1 | 1
Not completed — Other, Not Specified | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received any dose of study drug, analyzed according to the treatment randomized.
Groups:
- Placebo: Participants received IV infusion of placebo matched to VIB4920 on Days 1, 15, 29, and 57.
- Total: Total of all reporting groups
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times | Total
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 15 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (14.0) | 53.2 (10.7) | 59.0 (12.2) | 56.5 (12.2) | 56.4 (15.2) | 56.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 11 | 13 | 12 | 62
  Male | 4 | 2 | 5 | 2 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 15 | 15 | 15 | 15 | 15 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 0 | 1 | 1 | 4
  White | 14 | 16 | 15 | 14 | 14 | 73
  Other, Not Specified | 0 | 0 | 1 | 0 | 0 | 1
Disease Activity Score 28 C-reactive Protein (DAS28-CRP) [Mean (Standard Deviation); unit: score on a scale] — The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity.
  score on a scale | 5.443 (1.066) | 5.473 (0.883) | 5.945 (0.736) | 5.452 (0.644) | 5.761 (0.711) | 5.615 (0.830)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 113 in DAS28-CRP
Description: The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from baseline indicates improvement in disease activity. Results are from a mixed-effect model for repeated measures (MMRM) analysis with treatment, visit, visit by treatment interaction, and baseline DAS28-CRP score included in the model.
Time Frame: Day 1 (Baseline), Day 113
Population: Full Analysis Set: all randomized participants who received any dose of study drug, analyzed according to the treatment randomized. Participants with an assessment at given time point by group.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 15 | 14 | 15 | 14 | 14
score on a scale | -1.06 (0.26) | -1.90 (0.27) | -1.87 (0.27) | -1.87 (0.27) | -1.83 (0.28)
Statistical Analysis 1: Comparison: Placebo vs VIB4920 3000 mg Once; Test type: Superiority; p = 0.0296, MMRM — Results are from MMRM analysis with treatment, visit, visit by treatment interaction, and baseline DAS28-CRP score included in the model; Least Squares (LS) Mean Difference = -0.84, 90% CI 2-sided [-1.47 to -0.21], Standard Error of Mean 0.38 — LS Mean difference is VIB4920 minus placebo. Differences less than 0 favor VIB4920
Statistical Analysis 2: Comparison: Placebo vs VIB4920 1500 mg Twice; Test type: Superiority; p = 0.0355, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.81, 90% CI 2-sided [-1.44 to -0.18], Standard Error of Mean 0.38 — LS Mean difference is VIB4920 minus placebo. Differences less than 0 favor VIB4920
Statistical Analysis 3: Comparison: Placebo vs VIB4920 3000 mg Twice; Test type: Superiority; p = 0.0364, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.81, 90% CI 2-sided [-1.44 to -0.18], Standard Error of Mean 0.38 — LS Mean difference is VIB4920 minus placebo. Differences less than 0 favor VIB4920
Statistical Analysis 4: Comparison: Placebo vs VIB4920 1500 mg 4 Times; Test type: Superiority; p = 0.0478, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.77, 90% CI 2-sided [-1.41 to -0.13], Standard Error of Mean 0.38 — LS Mean difference is VIB4920 minus placebo. Differences less than 0 favor VIB4920

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), and Treatment-emergent Adverse Events of Special Interest (TEAESIs)
Description: Adverse event (AE): any untoward medical occurrence associated with the use of an intervention in humans, whether or not it is considered intervention-related. Serious adverse event (SAE): an AE that results in any of the following outcomes: death; life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity; congenital anomaly/birth defect; other important medical event jeopardizing the participant's well-being. AEs of special interest (AESIs) include: thrombotic and embolic events; anaphylaxis and clinically significant (Common Terminology Criteria for Adverse Events [CTCAE] Grade 3 or higher) hypersensitivity reactions; severe infusion-related reactions (CTCAE Grade 3 or higher); immune complex disease; severe (CTCAE Grade 3 or higher) and/or opportunistic infections; hepatic function abnormality meeting the definition of Hy's Law; malignant neoplasm. (CTCAE Grade 3=Severe; Grade 4=Life-threatening; Grade 5=Fatal.)
Time Frame: From first dose of study drug through Day 309 ± 7 days
Population: Safety analysis set: all participants who received any dose of study drug, analyzed according to the treatment that they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 18 | 17 | 13 | 14
Participants
  At least one event | 10 | 10 | 14 | 11 | 11
  At least one study drug-related event | 4 | 3 | 4 | 2 | 2
  At least one event of ≥ Grade 3 severity | 0 | 1 | 1 | 0 | 0
  Death (Grade 5 severity) | 0 | 0 | 1 | 0 | 0
  At least one serious event | 0 | 1 | 1 | 0 | 1
  At least one serious and/or ≥ Grade 3 severity event | 0 | 1 | 1 | 0 | 0
  At least one related serious event | 0 | 0 | 0 | 0 | 0
  At least one event leading to discontinuation of study drug | 0 | 1 | 0 | 0 | 0
  At least one event of special interest | 0 | 1 | 1 | 0 | 0

3. Secondary Outcome: Pharmacokinetics (PK) of VIB4920: Maximum Observed Concentration (Cmax)
Time Frame: Predose (within 30 minutes prior to start of infusion), and within 10 minutes of the end of infusion on Days 1 (Dose 1), 15 ± 1 day (d; Dose 2), 29 ± 3d (Dose 3), 57 ± 3d (Dose 4), and Days 85 ± 3d, 113 ± 5d, 141 ± 5d, 169 ± 5d, 197 ± 7d, 225 ± 7d
Population: PK Analysis Set: Participants who received active study drug and had at least one quantifiable plasma PK observation post-first dose. Participants were analyzed according to the treatment that they actually received. Participants with an assessment at given dose time points by group.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 17 | 13 | 14
μg/mL
  Dose 1: number analyzed (Participants) | 16 | 17 | 13 | 13
  Dose 1 | 877 (204) | 476 (127) | 860 (275) | 421 (102)
  Dose 2: number analyzed (Participants) | 0 | 15 | 13 | 13
  Dose 2 |  | 504 (162) | 1050 (349) | 564 (163)
  Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 3 |  |  |  | 601 (181)
  Dose 4: number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 4 |  |  |  | 568 (140)

4. Secondary Outcome: PK of VIB4920: Time to Cmax (Tmax)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: day
Arm/Group | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 17 | 13 | 14
day
  Dose 1: number analyzed (Participants) | 16 | 17 | 13 | 13
  Dose 1 | 0.0899 [0.0868 to 0.100] | 0.0875 [0.0847 to 0.0951] | 0.0875 [0.0840 to 0.0917] | 0.0903 [0.0840 to 0.108]
  Dose 2: number analyzed (Participants) | 0 | 15 | 13 | 13
  Dose 2 |  | 0.0681 [0.0646 to 0.0847] | 0.0667 [0.0486 to 0.0882] | 0.0486 [0.0437 to 0.0521]
  Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 3 |  |  |  | 0.0472 [0.0438 to 0.0486]
  Dose 4: number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 4 |  |  |  | 0.0667 [0.0486 to 0.0708]

5. Secondary Outcome: PK of VIB4920: Area Under the Concentration-Time Curve From Time 0 to the Last Quantifiable Concentration (AUClast)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μg·day/mL
Arm/Group | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 17 | 13 | 14
μg·day/mL
  Dose 1: number analyzed (Participants) | 16 | 17 | 13 | 13
  Dose 1 | 7350 (1380) | 3980 (1580) | 7870 (2570) | 2960 (604)
  Dose 2: number analyzed (Participants) | 0 | 15 | 13 | 13
  Dose 2 |  | 5280 (2000) | 10000 (3320) | 4060 (1290)
  Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 3 |  |  |  | 6350 (1840)
  Dose 4: number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 4 |  |  |  | 5770 (1110)

6. Secondary Outcome: PK of VIB4920: Area Under the Concentration-Time Curve From Time 0 to Day 56 (AUC0-56D)
Time Frame: Predose (within 30 minutes prior to start of infusion), and within 10 minutes of the end of infusion on Days 1 (Dose 1), 15 ± 1 day (d; Dose 2), 29 ± 3d (Dose 3), Day 56
Population: PK Analysis Set: Participants who received active study drug and had at least one quantifiable plasma PK observation post-first dose. Participants were analyzed according to the treatment that they actually received. Participants with an assessment at given dose time points by group. Per protocol, due to the nature of the dosing and sampling for the VIB4920 1500 mg 4 Times arm, this analysis was not done.
Measure: Mean (Standard Deviation); unit: μg·day/mL
Arm/Group | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 15 | 13 | 0
μg·day/mL
  Dose 1 | 7280 (1370) | 4280 (1280) | 7870 (2570) |
  Dose 2: number analyzed (Participants) | 0 | 14 | 13 | 0
  Dose 2 |  | 5310 (2000) | 9910 (3250) |
  Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Dose 4: number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: PK of VIB4920: Total Body Clearance (CL) for Dose 1 and Total Body Clearance at Steady State (CLss) for Doses 2 to 4
Time Frame: as for outcome 3
Population: PK Analysis Set: Participants who received active study drug and had at least one quantifiable plasma PK observation post-first dose. Participants were analyzed according to the treatment that they actually received. Participants with an assessment at given dose time points by group. Per protocol, due to the nature of the dosing and sampling for the VIB4920 1500 mg 4 Times arm, this analysis was done for Dose 4 only.
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 15 | 15 | 13 | 14
mL/day
  Dose 1 (CL): number analyzed (Participants) | 15 | 15 | 13 | 0
  Dose 1 (CL) | 430 (91.9) | 371 (92.5) | 417 (144) |
  Dose 2 (CLss): number analyzed (Participants) | 0 | 14 | 13 | 0
  Dose 2 (CLss) |  | 314 (104) | 340 (140) |
  Dose 3 (CLss): number analyzed (Participants) | 0 | 0 | 0 | 0
  Dose 4 (CLss): number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 4 (CLss) |  |  |  | 294 (49.8)

8. Secondary Outcome: PK of VIB4920: Terminal Elimination Half-Life (t1/2)
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: day
Arm/Group | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 15 | 13 | 14
day
  Dose 1: number analyzed (Participants) | 16 | 15 | 13 | 0
  Dose 1 | 9.27 (1.61) | 9.06 (1.98) | 9.02 (1.06) |
  Dose 2: number analyzed (Participants) | 0 | 14 | 13 | 0
  Dose 2 |  | 9.55 (1.51) | 9.88 (1.41) |
  Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Dose 4: number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 4 |  |  |  | 10.5 (2.06)

9. Secondary Outcome: PK of VIB4920: Volume of Distribution at Steady State (Vss)
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 15 | 15 | 13 | 14
mL
  Dose 1: number analyzed (Participants) | 15 | 15 | 13 | 0
  Dose 1 | 4350 (1300) | 3750 (601) | 4540 (1470) |
  Dose 2: number analyzed (Participants) | 0 | 14 | 13 | 0
  Dose 2 |  | 3490 (926) | 3600 (1720) |
  Dose 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Dose 4: number analyzed (Participants) | 0 | 0 | 0 | 14
  Dose 4 |  |  |  | 3210 (865)

10. Secondary Outcome: Total Soluble Cluster of Differentiation 40 Ligand (sCD40L) Plasma Concentration Over Time
Description: Total sCD40L (free sCD40L and sCD40L bound to VIB4920) was measured in plasma samples using a modified commercially available kit.
Time Frame: Day 1 (Baseline), Days 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 15
ng/mL
  Change at Day 15: number analyzed (Participants) | 16 | 16 | 16 | 13 | 14
  Change at Day 15 | 4.6759 (3.6596) | 30.7744 (7.4954) | 36.0088 (14.4324) | 28.2492 (10.4252) | 33.9007 (8.7777)
  Change at Day 29: number analyzed (Participants) | 16 | 15 | 15 | 14 | 14
  Change at Day 29 | 4.8431 (3.3770) | 67.5427 (16.4322) | 66.7047 (15.3708) | 68.0636 (28.6523) | 68.1386 (12.1314)
  Change at Day 57: number analyzed (Participants) | 16 | 15 | 15 | 14 | 14
  Change at Day 57 | 0.8150 (1.6053) | 64.4177 (16.4322) | 62.5560 (14.4445) | 63.6939 (25.5500) | 64.1329 (12.4842)
  Change at Day 85: number analyzed (Participants) | 15 | 15 | 15 | 15 | 14
  Change at Day 85 | 0.4483 (1.1842) | 53.1583 (20.6513) | 77.5360 (18.7440) | 57.2587 (20.0742) | 69.8821 (19.2623)
  Change at Day 113: number analyzed (Participants) | 15 | 14 | 15 | 14 | 14
  Change at Day 113 | 0.3420 (1.3246) | 21.4686 (19.3705) | 75.4407 (18.2921) | 53.4514 (26.2712) | 68.5636 (19.3458)
  Change at Day 141: number analyzed (Participants) | 15 | 15 | 14 | 15 | 14
  Change at Day 141 | 0.2547 (0.9863) | 1.6517 (3.7565) | 55.4204 (28.9470) | 53.2827 (31.6165) | 52.3943 (29.4422)
  Change at Day 169: number analyzed (Participants) | 14 | 15 | 14 | 15 | 13
  Change at Day 169 | 0.3114 (1.1653) | 0 (0) | 21.1296 (27.1973) | 18.3170 (20.2842) | 23.5727 (26.0510)
  Change at Day 197: number analyzed (Participants) | 14 | 14 | 14 | 15 | 14
  Change at Day 197 | 0.2757 (1.0316) | 0 (0) | 4.4354 (9.9146) | 2.5057 (4.4880) | 4.6343 (5.3603)
  Change at Day 225: number analyzed (Participants) | 14 | 14 | 14 | 15 | 14
  Change at Day 225 | 0.2450 (0.9167) | 0 (0) | -0.4043 (1.5127) | -0.0137 (1.1940) | -0.2971 (0.8718)
  Change at Day 253: number analyzed (Participants) | 14 | 14 | 13 | 13 | 13
  Change at Day 253 | 0.3436 (1.2855) | 3.1418 (11.7555) | -0.5946 (2.1439) | -0.5292 (1.9082) | -0.9485 (2.3281)
  Change at Day 281: number analyzed (Participants) | 14 | 13 | 10 | 14 | 13
  Change at Day 281 | -0.0343 (0.1283) | 0 (0) | -0.5640 (1.7835) | -0.4729 (1.7693) | -0.9485 (2.3281)
  Change at Day 309: number analyzed (Participants) | 14 | 12 | 10 | 12 | 13
  Change at Day 309 | -0.5654 (2.1154) | 0 (0) | -0.5720 (1.8088) | -0.7833 (2.7135) | -0.9485 (2.3281)

11. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibodies (ADA) to VIB4920
Description: ADA positive at any time: observed at least once during the study (baseline included).
  Treatment-emergent ADA: ADA positive post-baseline only or boosted pre-existing ADA during the study period.
  Persistent positive: treatment-induced ADA positive at ≥ 2 post-baseline assessments (with ≥ 16 weeks between first and last positive) or positive at last post-baseline assessment.
  Transient positive: treatment-induced ADA post-baseline positive but does not fulfill the criteria of persistent positive.
Time Frame: Day 1 (Baseline) to Day 309 Day 1 (Baseline) up to Day 309 (± 7 days)
Population: Safety analysis set: all participants who received any dose of study drug, analyzed according to the treatment that they actually received. Participants who received active study drug.
Measure: Number; unit: percentage of participants
Arm/Group | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 18 | 17 | 13 | 14
percentage of participants
  ADA positive at any time | 44.4 | 11.8 | 38.5 | 28.6
  Baseline ADA positive | 0 | 0 | 0 | 0
  Baseline only ADA positive | 0 | 0 | 0 | 0
  Post-baseline ADA positive | 44.4 | 11.8 | 38.5 | 28.6
  Treatment-emergent ADA | 44.4 | 11.8 | 38.5 | 28.6
  Persistent positive | 11.1 | 0 | 0 | 0
  Transient positive | 33.3 | 11.8 | 38.5 | 28.6

12. Secondary Outcome: Change From Baseline to Day 113 in Anti-Citrullinated Protein Antibodies (ACPAs)
Description: Excluding data after rescue. Adjusted geometric mean ratio to baseline (90% CI) results are from MMRM analysis on log(ratio to baseline) with treatment, visit, visit by treatment interaction, and log(baseline) included in the model. Ratios less than 1 indicate a decrease.
Time Frame: Day 1 (Baseline), Day 113
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 15 | 14 | 15 | 14 | 14
ratio | 1.08 [0.83 to 1.42] | 0.69 [0.52 to 0.91] | 0.82 [0.62 to 1.07] | 0.84 [0.63 to 1.11] | 0.62 [0.47 to 0.82]
Statistical Analysis 1: Comparison: Placebo vs VIB4920 3000 mg Once; Test type: Superiority; p = 0.0584, MMRM — Results are from MMRM analysis on log(ratio to baseline) with treatment, visit, visit by treatment interaction, and log(baseline) included in the model; Ratio of geometric mean versus placebo = 0.64, 90% CI 2-sided [0.43 to 0.94] — Ratio of geometric mean is for VIB4920:placebo. Ratios less than 1 indicate a decrease
Statistical Analysis 2: Comparison: Placebo vs VIB4920 1500 mg Twice; Test type: Other; p = 0.2274, MMRM — [p-value comment as in outcome 12, analysis 1]; Ratio of geometric mean versus placebo = 0.76, 90% CI 2-sided [0.51 to 1.11] — Ratio of geometric mean is for VIB4920:placebo. Ratios less than 1 indicate a decrease
Statistical Analysis 3: Comparison: Placebo vs VIB4920 3000 mg Twice; Test type: Superiority; p = 0.2794, MMRM — [p-value comment as in outcome 12, analysis 1]; Ratio of geometric mean versus placebo = 0.77, 90% CI 2-sided [0.52 to 1.14] — Ratio of geometric mean is for VIB4920:placebo. Ratios less than 1 indicate a decrease
Statistical Analysis 4: Comparison: Placebo vs VIB4920 1500 mg 4 Times; Test type: Superiority; p = 0.0199, MMRM — [p-value comment as in outcome 12, analysis 1]; Ratio of geometric mean versus placebo = 0.57, 90% CI 2-sided [0.39 to 0.85] — Ratio of geometric mean is for VIB4920:placebo. Ratios less than 1 indicate a decrease

13. Secondary Outcome: Change From Baseline to Day 113 in Rheumatoid Factor (RF)
Description: as for outcome 12
Time Frame: Day 1 (Baseline), Day 113
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 15 | 14 | 15 | 14 | 14
ratio | 1.20 [1.04 to 1.39] | 0.77 [0.66 to 0.89] | 0.74 [0.64 to 0.86] | 0.72 [0.62 to 0.84] | 0.57 [0.49 to 0.66]
Statistical Analysis 1: Comparison: Placebo vs VIB4920 3000 mg Once; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 12, analysis 1]; Ratio of geometric mean versus placebo = 0.64, 90% CI 2-sided [0.52 to 0.79] — Ratio of geometric mean is for VIB4920:placebo. Ratios less than 1 indicate a decrease
Statistical Analysis 2: Comparison: Placebo vs VIB4920 1500 mg Twice; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 12, analysis 1]; Ratio of geometric mean versus placebo = 0.62, 90% CI 2-sided [0.50 to 0.76] — Ratio of geometric mean is for VIB4920:placebo. Ratios less than 1 indicate a decrease
Statistical Analysis 3: Comparison: Placebo vs VIB4920 3000 mg Twice; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 12, analysis 1]; Ratio of geometric mean versus placebo = 0.60, 90% CI 2-sided [0.48 to 0.74] — Ratio of geometric mean is for VIB4920:placebo. Ratios less than 1 indicate a decrease
Statistical Analysis 4: Comparison: Placebo vs VIB4920 1500 mg 4 Times; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 12, analysis 1]; Ratio of geometric mean versus placebo = 0.47, 90% CI 2-sided [0.38 to 0.59] — Ratio of geometric mean is for VIB4920:placebo. Ratios less than 1 indicate a decrease

14. Secondary Outcome: Percentage of Participants With Clinical Remission at Day 113
Description: Clinical remission is defined as DAS28-CRP < 2.6. The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity.
Time Frame: Day 113
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 15
percentage of participants | 18.8 | 18.8 | 6.3 | 13.3 | 13.3
Statistical Analysis 1: Comparison: Placebo vs VIB4920 3000 mg Once; Test type: Superiority; p = 0.7750, Regression, Logistic — Results are from logistic regression analysis with treatment and baseline DAS28-CRP score included in the model; Odds Ratio (OR) = 1.4, 90% CI 2-sided [0.2 to 8.0] — Odds ratio is VIB4920/placebo, with associated 90% CI and p-value. Odds ratios greater than 1 favor VIB4920
Statistical Analysis 2: Comparison: Placebo vs VIB4920 1500 mg Twice; Test type: Superiority; p = 0.6974, Regression, Logistic — Results are from logistic regression analysis with treatment and baseline DAS28-CRP score included in the model; Odds Ratio (OR) = 0.6, 90% CI 2-sided [0.1 to 5.5] — (Lower limit of 90% CI is < 0.1.) Odds ratio is VIB4920/placebo, with associated 90% CI and p-value. Odds ratios greater than 1 favor VIB4920
Statistical Analysis 3: Comparison: Placebo vs VIB4920 3000 mg Twice; Test type: Superiority; p = 0.9318, Regression, Logistic — Results are from logistic regression analysis with treatment and baseline DAS28-CRP score included in the model; Odds Ratio (OR) = 0.9, 90% CI 2-sided [0.1 to 5.7] — Odds ratio is VIB4920/placebo, with associated 90% CI and p-value. Odds ratios greater than 1 favor VIB4920
Statistical Analysis 4: Comparison: Placebo vs VIB4920 1500 mg 4 Times; Test type: Superiority; p = 0.9108, Regression, Logistic — Results are from logistic regression analysis with treatment and baseline DAS28-CRP score included in the model; Odds Ratio (OR) = 0.9, 90% CI 2-sided [0.2 to 5.1] — Odds ratio is VIB4920/placebo, with associated 90% CI and p-value. Odds ratios greater than 1 favor VIB4920

15. Secondary Outcome: Time to Start of New Treatment for Rheumatoid Arthritis (Rescue Medication)
Description: Based on Kaplan-Meier method.
Time Frame: Day 1 (Baseline) up to Day 309 (± 7 days)
Population: Full Analysis Set: all randomized participants who received any dose of study drug, analyzed according to the treatment randomized. Participants who received rescue medication.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 15
days | NA [NA to NA] — Not calculable due to small number of participants rescued. | NA [NA to NA] — Not calculable due to small number of participants rescued. | NA [NA to NA] — Not calculable due to small number of participants rescued. | NA [NA to NA] — Not calculable due to small number of participants rescued. | NA [196 to NA] — Not calculable due to small number of participants rescued.
Statistical Analysis 1: Comparison: Placebo vs VIB4920 3000 mg Once; Test type: Superiority; p = 0.9805, Regression, Cox — Based on Cox regression method with treatment group included in the model; Hazard Ratio (HR) = 1.04, 90% CI 2-sided [0.10 to 10.60] — Hazard ratio is VIB4920/placebo. Hazard ratios less than 1 favor VIB4920
Statistical Analysis 2: Comparison: Placebo vs VIB4920 1500 mg Twice; Test type: Superiority; p = 0.9805, Regression, Cox — Based on Cox regression method with treatment group included in the model; Hazard Ratio (HR) = 1.04, 90% CI 2-sided [0.10 to 10.60] — Hazard ratio is VIB4920/placebo. Hazard ratios less than 1 favor VIB4920
Statistical Analysis 3: Comparison: Placebo vs VIB4920 3000 mg Twice; Test type: Superiority; p = 0.3407, Regression, Cox — Based on Cox regression method with treatment group included in the model; Hazard Ratio (HR) = 3.01, 90% CI 2-sided [0.45 to 20.09] — Hazard ratio is VIB4920/placebo. Hazard ratios less than 1 favor VIB4920
Statistical Analysis 4: Comparison: Placebo vs VIB4920 1500 mg 4 Times; Test type: Superiority; p = 0.9805, Regression, Cox — Based on Cox regression method with treatment group included in the model; Hazard Ratio (HR) = 1.04, 90% CI 2-sided [0.10 to 10.60] — Hazard ratio is VIB4920/placebo. Hazard ratios less than 1 favor VIB4920

ADVERSE EVENTS:
Time Frame: From screening (all cause mortality) or first dose of study drug (adverse events) through through Day 309 ± 7 days.
Description: Safety analysis set: all participants who received any dose of study drug, analyzed according to the treatment that they actually received.
Arm/Group | Placebo | VIB4920 3000 mg Once | VIB4920 1500 mg Twice | VIB4920 3000 mg Twice | VIB4920 1500 mg 4 Times
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18 | 1/17 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/18 | 1/17 | 0/13 | 1/14
Other Adverse Events (participants affected / at risk) | 10/16 | 10/18 | 14/17 | 11/13 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | VIB4920 3000 mg Once (N=18) | VIB4920 1500 mg Twice (N=17) | VIB4920 3000 mg Twice (N=13) | VIB4920 1500 mg 4 Times (N=14)
Death (General disorders) | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | VIB4920 3000 mg Once (N=18) | VIB4920 1500 mg Twice (N=17) | VIB4920 3000 mg Twice (N=13) | VIB4920 1500 mg 4 Times (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 3 | 0 | 3
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasal herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0
Blood glucose abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0
Heart sounds abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 antibody test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2 | 1
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Parkinsonian rest tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoid operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04163991/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04163991/SAP_001.pdf